CLINICAL TRIAL: NCT07112001
Title: Adaptation and Implementation of a Behavioral mHealth Intervention to Reduce Anxiety and Depression and End the HIV Epidemic in the Rural South
Brief Title: A Behavioral mHealth Intervention for People With HIV With Anxiety and Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 202003223; K23MH131463 (NIH)
Record Dates: First submitted 2025-07-22; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: HIV; Depression; Anxiety
Keywords: HIV; Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Counseling; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified PositiveLinks app with CHW-delivered counseling (Experimental): This arm includes a modified version of the PositiveLinks app which includes access to community health worker-delivered positive affect counseling via a video call feature on the app
  Interventions: Behavioral: PositiveLinks with Counseling
- Unmodified PositiveLinks with no counseling (Active Comparator): This arm includes the standard of care which includes the standard version of the PositiveLinks app and feedback on self-reported anxiety and depression symptoms and a list of local mental health resources
  Interventions: Behavioral: Standard of Care (SOC)

INTERVENTIONS:
Behavioral: PositiveLinks with Counseling — A community health worker delivered, specialized counseling intervention through video call on the PositiveLinks app
  Arms: Modified PositiveLinks app with CHW-delivered counseling
Behavioral: Standard of Care (SOC) — This intervention includes the use of the unmodified PositiveLinks app and the standard of care for addressing anxiety and depression in the HIV clinic
  Arms: Unmodified PositiveLinks with no counseling

SUMMARY:
This study will adapt and assess the preliminary effectiveness of a community health worker-delivered mental health counselling intervention delivered remotely to reduce anxiety and depression among people with HIV in Florida.

DETAILED DESCRIPTION:
The investigators will conduct a pilot randomized controlled trial to evaluate the preliminary effectiveness of an adapted community health worker (CWH)-delivered positive affect counselling intervention delivered remotely via mHealth. The adapted intervention will include CHW-delivered positive affect skill-based counseling accessible through video call that will be accessible through the mHealth app. The CHW will conduct approximately 5 weekly individual 60-minute counseling sessions via a secure video call feature. If the participant does not have symptomatic improvement, the CHW will refer the participant to a licensed mental health professional. Participants will be randomized to receive access to the counselling intervention that also includes modified features of the mHealth app with increased mental health resources (intervention arm) or to current standard of mental health care that includes the unmodified version of the app (control arm). Participants allocated to the intervention arm will receive the counseling intervention approximately weekly for 5 weeks. The study will continue to abstract data from participants' EMR and mHealth app for approximately 6 months after enrollment. To assess preliminary effectiveness, the investigators will analyze differences by condition in anxiety and depression (primary outcome). Informed consent will be obtained prior to study participation.

ELIGIBILITY:
Inclusion Criteria:

* HIV diagnosis
* GAD-7 score of 5 or greater
* PHQ-8 score of 5 or greater

Exclusion Criteria:

* Active psychosis
* Suicidal ideation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Reduction in Depression | 3 months
  The intervention aims to reduce depression. This will be assessed using the Patient Health Questionnaire-8 (PHQ-8). The minimum score is 0. The maximum score is 24. A higher score indicates a worse outcome.
Reduction in Anxiety | 3 months
  The intervention aims to reduce anxiety. This will be assessed using the Generalized Anxiety Disorder-7 (GAD-7). The minimum score is 0. The maximum score is 21. A higher score indicates a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD